CLINICAL TRIAL: NCT06018324
Title: CloudCare Patient Reported Outcomes in the Treatment of Type 1 Diabetes in Pediatrics A Prospective Cohort Study in Europe
Brief Title: CloudCare in the Treatment of Type 1 Diabetes in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diabeter Nederland BV (Other)
Responsible Party: Sponsor
Other Study IDs: DIA-2023-01
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Type1diabetes; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study aims to estimate the effect of the CloudCare application in daily practice on treatment satisfaction and emotional burden for pediatric patients and their parents/caregivers, patients' glycemic control (glucometrics), healthcare professional satisfaction, and the impact on costs.

A total of 600 pediatric patients (1-15 years) with type 1 diabetes will be enrolled into the study.

DETAILED DESCRIPTION:
This is a multi center prospective cohort study in Europe with pre- and post-measurements in type 1 diabetes with 12 months follow-up. This study will only include pediatric patients for which CloudCare is part of their (new) standard care of type 1 diabetes. Participants will be enrolled in several hospitals/healthcare organisations in Europe. Participant's data will be retrieved from their medical records and from uploaded data of their medical devices used for their type 1 diabetes treatment.

The study will consist of two periods. A 3 months' retrospective period in which data will be retrieved from patients' dossier followed by a 12 months' prospective period after introduction of CloudCare as part of patients' standard care by the treating physician.

The 3 months' retrospective period is the control period for the prospective period.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers and, depending on local laws and regulations, also the patient are willing to sign the study informed consent form prior to any data collection for this study
* Clinical diagnosis, based on investigator assessment, of type 1 diabetes and using insulin with or without metformin for at least 6 months.
* Age between 1 and 15 years old.
* Use of multiple daily injections of insulin (MDI, with a basal insulin injection and bolus injections) or continuous subcutaneous insulin infusion (CSII) with Flash or Continuous Glucose Monitoring (FGM/CGM), but without CloudCare for at least three months.
* Receiving CloudCare as part of their standard care for at least 6 months.

Exclusion Criteria:

* Patients with type 1 diabetes on glucose lowering treatments other than insulin with or without metformin.
* Any known factor, condition, or disease that might interfere with study conduct or interpretation of the results, as deemed by the investigator.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with type 1 diabetes (1-15 years). All participants must be treated with multiple daily injections of insulin (MDI) or continuous subcutaneous insulin infusion (CSII) with continuous or flash glucose monitoring (CGM/FGM) for at least three months without CloudCare and will get CloudCare as part of their standard care.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
DTSQc | 6 months
  Change in mean treatment satisfaction score at 6 months using change version of the Diabetes Treatment Satisfaction Questionnaire (DTSQc) for Teens and Parents

SECONDARY OUTCOMES:
DTSQs | 0, 6, 12 months
  Change in mean treatment satisfaction score at 0- 6- and 12-months using status version of the Diabetes Treatment Satisfaction Questionnaire (DTSQs) for Teens and Parents
Change in mean % HbA1c | -3 months to 3, 6 and 12 months
Change in mean TIR | -3 months to 3, 6 and 12 months
  Time in Range
Change in mean TAR | -3 months to 3, 6 and 12 months
  Time Above Range
Change in mean TBR | -3 months to 3, 6 and 12 months
  Time Below Range
Change in mean PAID-teens and PAID-parent | 0, 3, 6 and 12 months
Change in mean QoL score and mean QoL diabetes related score | 0, 3, 6 and 12 months
  Quality of Life; 2 questions
Change in mean treatment satisfaction score of the HCP satisfaction Questionnaire | 0, 3, 6 and 12 months
  Non-validated satisfaction questionnaire
Treatment costs | 0, 3, 6 and 12 months
  * Treatment costs of complications requiring hospitalizations
  * Number of contacts with HCP
  * Type of contacts with HCP (Face to face, Email/Telephone)
  * Time spent by the HCP

CONTACTS AND LOCATIONS:
Locations (1):
- Diabeter, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided